CLINICAL TRIAL: NCT01970306
Title: A Prospective Phase II Trial to Evaluate Esophageal Reinforcement With ACell MatriStem Surgical Matrix: A Degradable Biologic Scaffold Material
Brief Title: Evaluate Esophageal Reinforcement With ACell MatriStem Surgical Matrix: A Degradable Biologic Scaffold Material
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-178
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Adenocarcinoma
Keywords: Esophageal Reinforcement; ACell MatriStem; 13-178
MeSH Terms: conditions — Adenocarcinoma Of Esophagus

ARMS (1):
- Surgical intervention (Experimental): Patients will undergo standard resection and gastrointestinal anastomosis and will then have reinforcement of the anastomosis with MatriStem PSM. Patients undergoing esophagectomy, PG or TG will be evaluated with one routine postoperative contrast swallow study at post-operative day #4-10.
  Interventions: Device: MatriStem PSM

INTERVENTIONS:
Device: MatriStem PSM — All esophageal anastomoses will be reinforced circumferentially with ACell MatriStem PSM.

SUMMARY:
The purpose of this study is to see if implanting MatriStem will lower the risk of one of the more common complications after stomach or esophagus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Pathologically confirmed Gastric, Gastroesophageal Junction (GEJ) or Esophageal, adenocarcinoma at either MSKCC or a participating site (biopsy may be performed at other institutions but slides must be confirmed at MSKCC or a participating site, as is routine care at our institution)
* Patient undergoing any resection requiring an anastomosis to the esophagus for curative intent. Including but not limited to esophagectomy or total gastrectomy.
* Subject is willing to provide written informed consent
* Subject is willing and able to comply with the follow-up regimen

Exclusion Criteria:

* Pregnant or lactating women
* Intraoperative evidence of metastatic or locally-unresectable disease
* Patients with known sensitivity or allergy to porcine materials.
* Patients undergoing any resection requiring an anastomosis to the esophagus for palliative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Strong, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Vos EL, Nakauchi M, Capanu M, Park BJ, Coit DG, Molena D, Yoon SS, Jones DR, Strong VE. Phase II Trial Evaluating Esophageal Anastomotic Reinforcement with a Biologic, Degradable, Extracellular Matrix after Total Gastrectomy and Esophagectomy. J Am Coll Surg. 2022 May 1;234(5):910-917. doi: 10.1097/XCS.0000000000000113. PMID 35426405
- [Derived] Shannon AB, Straker RJ 3rd, Fraker DL, Miura JT, Karakousis GC. Validated Risk-Score Model Predicting Lymph Node Metastases in Patients with Non-Functional Gastroenteropancreatic Neuroendocrine Tumors. J Am Coll Surg. 2022 May 1;234(5):900-909. doi: 10.1097/XCS.0000000000000144. PMID 35426404
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgical Intervention: Patients will undergo standard resection and gastrointestinal anastomosis and will then have reinforcement of the anastomosis with MatriStem PSM.
Period: Overall Study
Arm/Group | Surgical Intervention
Started | 78
Completed | 66
Not Completed | 12
Not completed — Not eligible | 3
Not completed — Not able to be treated | 9

BASELINE CHARACTERISTICS:
Arm/Group | Surgical Intervention
Number analyzed (Participants) | 78
Age, Continuous [Median (Full Range); unit: years] | 66 [21 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 67
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anastomotic Leak.
Description: Anastomotic leak will be assessed by clinical observation and one postoperative contrast study (thin-barium Gastrografin or Omnipaque swallow)
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Intervention
Number analyzed (Participants) | 78
Participants
  Participants diagnosed with anastomotic leak | 10
  Participants without anastomotic leak | 68

2. Secondary Outcome: Stricture Formation Clinically and by Determination of Dysphagia Score
Description: Patients will be evaluated in the outpatient clinic and will be assigned a dysphagia score from 0-4 by the RSA. Patients reporting symptoms consistent with stricture will be evaluated with radiographic contrast swallow study or endoscopy.
Time Frame: 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Intervention
Number analyzed (Participants) | 78
Participants
  Not evaluable | 14
  No reported dysphagia | 54
  Dysphagia | 10

3. Secondary Outcome: Number of Participants Who Developed Anastomotic Stenosis
Description: If during the follow up period, patients report any symptoms suggestive of anastomotic stricture, a contrast study (esophagram) or endoscopy will be obtained at that time to evaluate for stricture. These tests will be performed as per standard postoperative assessment by the surgeon.
Time Frame: 90 days post op
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Intervention
Number analyzed (Participants) | 78
Participants
  Not evaluable | 14
  Anastomotic stenosis | 8
  No anastomotic stenosis | 56

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Surgical Intervention
All-Cause Mortality (participants affected / at risk) | 29/78
Serious Adverse Events (participants affected / at risk) | 18/78
Other Adverse Events (participants affected / at risk) | 8/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgical Intervention (N=78)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Death NOS (General disorders) | 1
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 7
Esophageal stenosis (Gastrointestinal disorders) | 3
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 1
Gastric necrosis (Gastrointestinal disorders) | 1
Heart failure (Cardiac disorders) | 1
Hepatic infection (Infections and infestations) | 1
Ileus (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgical Intervention (N=78)
Stomach pain (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT01970306/Prot_SAP_000.pdf